CLINICAL TRIAL: NCT05708833
Title: Intra-Osseous Access in Difficult Vascular Access Cases
Acronym: IODA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P170918J
Record Dates: First submitted 2022-04-06; First posted 2023-02-01 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Hemodynamic Instability

STUDY DESIGN:
Intervention Model Description: Interventional study with randomisation (1:1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intraosseous venous access (Experimental): intraosseous venous access
  Interventions: Device: Intraosseous venous access
- peripheral venous access (Active Comparator): Limiting use of intraosseous access (intraosseous access possible after 3 attempts of peripheral venous access)
  Interventions: Device: Peripheral venous access

INTERVENTIONS:
Device: Intraosseous venous access — Immediate placement of humeral intra-osseous venous access (after a first failed attempt of peripheral venous access)
  Arms: intraosseous venous access
Device: Peripheral venous access — Looking for peripheral venous access, changing the site of puncture, the caliber of the catheter and/or the operator and/or assistance tools (ultrasound, infra-red guidance...) and/or using another route (oral, rectal, subcutaneous, intramuscular route and central venous access)
  Arms: peripheral venous access

SUMMARY:
Thousands of peripheral venous accesses are inserted every day all over the world. Some of them, such as those inserted in emergency and / or in critical patients, are absolutely vital. In the particular context of prehospital care, the rate of failure of the first attempt to insert a peripheral venous access has been evaluated at 25%. Success rates of successive attempts were about 75%. Nevertheless, the final success rate is close to 100%.

Failure or delay in obtaining venous access can be life-threatening. Thus, alternatives to peripheral venous access have been proposed including intraosseous route recently made easier by the development of an automated puncture device (EZ-IO®), but still rarely used, especially on conscious patient.

Currently, the place of intraosseous venous access in critical patients is not determined.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient, in prehospital setting, without venous access and after failure of the first attempt to place a peripheral venous access by a senior operator (doctor or nurse) AND
2. Patient with hemodynamic failure defined as:

   * systolic blood pressure (SBP) < 90 mm Hg (2 measures) or
   * cardiac arrest or
3. Any situation requiring intubation

Exclusion Criteria:

* 1- Age < 18 years

  2- Venous access already available

  3- Known contra-indications to intraosseous access (i.e. bilateral lesions):
* Bone fracture
* Skin infection
* Osteoporosis
* Osteomyelitis
* Local burns
* Recent failed intraosseous attempt
* Prior surgery
* Compartment syndrome
* Every other local specific situations

  4- Pregnancy woman

  5- Patient with no national health or universal plan affiliation coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
To demonstrate that the early recourse to the intraosseous route, from the first failure, makes it possible to obtain more quickly the correction of the failure of critical patient managed in prehospital setting. | • In patients with cardiac arrest: Return of spontaneous circulation (ROSC), an average of 1 hour
  • In patients with cardiac arrest: Time required for a return of spontaneous circulation (ROSC).
  Only the first ROSC will be considered.
To demonstrate that the early recourse to the intraosseous route, from the first failure, makes it possible to obtain more quickly the correction of the failure of critical patient managed in prehospital setting. | • In patients with hemodynamic failure: Reach a systolic blood pressure correction, an average of 1 hour
  • In patients with hemodynamic failure: delay to reach a systolic blood pressure correction, i.e. systolic blood pressure > 90 mm Hg.
  Systolic blood pressure will be assessed every 5 minutes after the placement of the intravenous line. Two consecutive measures are required to reach the end-point.
  In the cases where continuous invasive blood pressure monitoring will be available, systolic blood pressure > 90 mm Hg > 1 minute will be required.
To demonstrate that the early recourse to the intraosseous route, from the first failure, makes it possible to obtain more quickly the correction of the failure of critical patient managed in prehospital setting. | • In patients requiring endo-tracheal intubation: Achieve intubation, an average of 1 hour
  • In patients requiring endo-tracheal intubation: time required to achieve intubation.

SECONDARY OUTCOMES:
To characterize the conditions for implementation of the procedure, depending on the strategy used. | 1 minute
  Failure to place the catheter defined by the absence of infusion or by withdrawal of the catheter within one minute after the opening of the infusion
To characterize the conditions for implementation of the procedure, depending on the strategy used. | In patients with cardiac arrest: Return of spontaneous circulation (ROSC), an average of 1 hour
  Number of punctures
To characterize the conditions for implementation of the procedure, depending on the strategy used. | In patients with hemodynamic failure: Reach a systolic blood pressure correction, an average of 1 hour
  Number of punctures
To characterize the conditions for implementation of the procedure, depending on the strategy used. | In patients requiring endo-tracheal intubation: Achieve intubation, an average of 1 hour
  Number of sites treated
To characterize the conditions for implementation of the procedure, depending on the strategy used. | In patients with cardiac arrest: Return of spontaneous circulation (ROSC). In patients with hemodynamic failure: Reach a systolic blood pressure correction. In patients requiring endo-tracheal intubation: Achieve intubation
  Use of alternative routes (central venous access, oral, rectal, subcutaneous, intramuscular - and intra-osseous in the control group)
To characterize the conditions for implementation of the procedure, depending on the strategy used. | In patients with cardiac arrest: Return of spontaneous circulation (ROSC), an average of 1 hour
  Use of alternative routes (central venous access, oral, rectal, subcutaneous, intramuscular - and intra-osseous in the control group)
To characterize the conditions for implementation of the procedure, depending on the strategy used. | In patients with hemodynamic failure: Reach a systolic blood pressure correction, an average of 1 hour
  Use of alternative routes (central venous access, oral, rectal, subcutaneous, intramuscular - and intra-osseous in the control group)
To characterize the conditions for implementation of the procedure, depending on the strategy used. | In patients requiring endo-tracheal intubation: Achieve intubation, an average of 1 hour
  Use of assistance tools (ultrasound, infra-red)
To characterize the conditions for implementation of the procedure, depending on the strategy used. | In patients with cardiac arrest: Return of spontaneous circulation (ROSC). In patients with hemodynamic failure: Reach a systolic blood pressure correction. In patients requiring endo-tracheal intubation: Achieve intubation
  Delays in placing venous access
To characterize the conditions for implementation of the procedure, depending on the strategy used. | In patients with cardiac arrest: Return of spontaneous circulation (ROSC), an average of 1 hour
  Delays in placing venous access
To characterize the conditions for implementation of the procedure, depending on the strategy used. | In patients with hemodynamic failure: Reach a systolic blood pressure correction, an average of 1 hour
  Delays in placing venous access
To characterize the conditions for implementation of the procedure, depending on the strategy used. | In patients with cardiac arrest: Return of spontaneous circulation (ROSC), an average of 1 hour
  Delays for administration of drugs/solutes
To characterize the conditions for implementation of the procedure, depending on the strategy used. | In patients with hemodynamic failure: Reach a systolic blood pressure correction, an average of 1 hour
  Delays for administration of drugs/solutes
To characterize the conditions for implementation of the procedure, depending on the strategy used. | In patients requiring endo-tracheal intubation: Achieve intubation, an average of 1 hour
  Delays for administration of drugs/solutes
To determine the length of stay in hospital | Days 28
  Length of stay in hospital
To evaluate morbidity depending on the strategy used. | In patients with cardiac arrest: Return of spontaneous circulation (ROSC), an average of 1 hour
  Non-functional venous
To evaluate morbidity depending on the strategy used. | In patients with hemodynamic failure: Reach a systolic blood pressure correction, an average of 1 hour
  Non-functional venous
To evaluate morbidity depending on the strategy used. | IIn patients requiring endo-tracheal intubation: Achieve intubation, In patients with hemodynamic failure: Reach a systolic blood pressure correction, an average of 1 hour
  Non-functional venous
To evaluate morbidity depending on the strategy used. | Days 28
  Local complication (subcutaneous diffusion, hematoma, pain...)
To evaluate morbidity depending on the strategy used. | Hours 72
  Need to replace the venous access
To evaluate mortality depending on the strategy used. | Days 28
  Death
To evaluate the patient's feedback, depending on the strategy used. | Immediately after the insertion of the catheter (opening of the perfusion) and on arrival at the hospital, In patients with hemodynamic failure: Reach a systolic blood pressure correction, an average of 1 hour
  Evaluation of procedural pain on an analog visual scale, EVA, simple verbal scale, EVS or numerical scale, EN (from 0 to 100, the higher is the worse) In the case of patient with cardiac arrest, only the operator satisfaction will be assessed.
To evaluate the team's feedback, depending on the strategy used. | Immediately after the insertion of the catheter (opening of the perfusion) and on arrival at the hospital, In patients with hemodynamic failure: Reach a systolic blood pressure correction, an average of 1 hour
  Operator satisfaction assessed (EVA, EVS or EN) after the placement of the catheter and on arrival at the hospital (from 0 to 100, the higher is the worse).

CONTACTS AND LOCATIONS:
Overall Officials: LAPOSTOLLE Frédéric, PhD MD, Principal Investigator — APHP
Locations (1):
- Hôpital Avicenne, Bobigny, France, France

IPD SHARING:
Plan to Share IPD: No